CLINICAL TRIAL: NCT05244434
Title: Comparative Effects of Ribociclib and Palbociclib on Circulating and Tumor Infiltrating Myeloid Cells in Metastatic Breast Cancer Patients
Brief Title: Effects of Ribociclib and Palbociclib on Tumor and Blood Characteristics in Patients With Metastatic Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI withdrawn
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21623; NCI-2022-00238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21623 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Advanced Breast Adenocarcinoma; Advanced HER2-Negative Breast Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Hormone Receptor-Positive Breast Carcinoma; Metastatic Breast Adenocarcinoma; Metastatic HER2-Negative Breast Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective cohort (SOC treatment, biopsy, blood collection) (Experimental): Patients receive SOC treatment consisting of ribociclib or palbociclib plus AI. Patients undergo biopsy of tumor tissue at baseline and post-treatment. Patients also undergo collection of blood samples at baseline, on day 1 of SOC treatment cycles 2, 4, and 6, every 6 cycles thereafter, and at post-treatment.
  Interventions: Other: Best Practice; Procedure: Biopsy; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis
- Retrospective cohort (Experimental): Patients' tumor tissue collected during previous SOC treatment (ribociclib or palbociclib plus AI) is used for analysis.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Best Practice — Given standard of care ribociclib + AI or palbociclib + AI
  Other Names: standard of care; standard therapy
  Arms: Prospective cohort (SOC treatment, biopsy, blood collection)
Procedure: Biopsy — Undergo biopsy of tumor tissue
  Other Names: BIOPSY_TYPE; Bx
  Arms: Prospective cohort (SOC treatment, biopsy, blood collection)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected
  Arms: Prospective cohort (SOC treatment, biopsy, blood collection)
Other: Laboratory Biomarker Analysis — Undergo analysis of previously collected tumor tissue

SUMMARY:
This clinical trial attempts to understand the differences between two chemotherapy drugs, ribociclib and palbociclib, and how they fight cancer. This study looks at tissue and blood characteristics of patients receiving these therapies in the hopes to develop a way to predict which medication would provide the most benefit to an individual patient.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify predictive immune biomarkers and mechanisms of response to ribociclib or palbociclib in advanced, hormone receptor positive breast cancer patients.

SECONDARY OBJECTIVES:

I. Identify changes in antigen presentation machinery and costimulatory molecules on circulating myeloid cells as a result of ribociclib or palbociclib treatment.

II. Characterize the dynamic remodeling of circulating myeloid cell composition that occur as a result of ribociclib or palbociclib treatment.

III. Characterize acquired immune tumor microenvironment features of resistance in patients that progress while undergoing ribociclib or palbociclib treatment.

EXPLORATORY OBJECTIVE:

I. To study the association between immune biomarkers and clinical response.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

PROSPECTIVE COHORT: Patients receive standard of care (SOC) treatment consisting of ribociclib or palbociclib plus aromatase inhibitor (AI). Patients undergo biopsy of tumor tissue at baseline and post-treatment. Patients also undergo collection of blood samples at baseline, on day 1 of SOC treatment cycles 2, 4, and 6, every 6 cycles thereafter, and at post-treatment.

RETROSPECTIVE COHORT: Patients' tumor tissue collected during previous SOC treatment (ribociclib or palbociclib plus AI) is used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmed breast adenocarcinoma who meet the following criteria:
* Age: >= 18 years and are post-menopausal
* Estrogen receptor positive (ER+) and human epidermal growth factor receptor 2 (HER2) negative breast cancer patients who prospectively may undergo evaluation for Cyclin-dependent kinase 4 and 6 inhibitors (CDK4/6i), ribociclib or palbociclib, as part of first-line therapy. Retrospective cohorts will be built to include either ribociclib or palbociclib treated patients with known clinical outcome
* During routine standard of care procedure, tumor that is accessible for ultrasound guided biopsy (from breast, lymph node, subcutaneous tumor, or selected liver metastasis per treating physician's discretion) or skin punch biopsy (for dermal metastasis) will be collected
* Available tumor tissue or planning on biopsy prior to initiation of CDK4/6i treatment
* Available tumor tissue or planning on biopsy at time of progression, prior to initiating subsequent therapy
* Willing to provide consent for extra tissue and blood samples

Exclusion Criteria:

* Patient received prior treatment with any CDK4/6 inhibitor
* Prior treatment with any chemotherapy for metastatic disease
* Patient is cognitively impaired
* Lung or bone metastasis only (not accessible by ultrasound guided biopsy)
* Patients with central nervous system (CNS) involvement unless they meet ALL the following criteria:

  * Untreated brain metastases (e.g., lesions < 1cm) not needing immediate local therapy
  * Previously treated brain metastases not needing immediate local therapy
  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment

    * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug:

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
  * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
  * Herbal preparations/medications, dietary supplements
  * Warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), newer anticoagulation agents such as direct factor Xa inhibitors, or fondaparinux is allowed
* Patient is currently receiving or has received systemic corticosteroids =< 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment

  * The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-03 (Estimated); Primary Completion 2023-01-26 (Estimated); Study Completion 2023-01-26 (Estimated)

PRIMARY OUTCOMES:
Immune cell frequency (relative abundance, cells per parental cell) | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Will be assessed by high dimensional flow cytometry. One-way analysis of variance (ANOVAs) and non-parametric Kruskal-Wallis tests will be used to compare relative abundances across patient groups and over the course of therapy. Wilcoxon rank-sum test will be used to examine the association between each biomarker of each sample collection and pathological response as appropriate. Odds ratios and 95% conference intervals will be calculated to measure strength of associations. P-values < 0.05 will be considered statistically significant. No adjustment for multiple comparisons will be used in view of the exploratory nature of this analysis.

SECONDARY OUTCOMES:
Single-cell gene expression | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Expected to identify > 30 myeloid and lymphocyte immune subsets. Gene expression relating to maturation and function will be focused on in myeloid subsets especially. Will be assessed by single-cell ribonucleic acid (RNA) sequencing. Immune cell type identification and gene expression patterns will be identified by unsupervised clustering and non-linear dimensionality reduction approaches. Cluster biomarkers will be identified by Seurat for annotating cell types (or functions) for each cell. Within each cluster, will compare the cellular differences in RNA expression across response and non-response cohorts of tumor and peripheral blood mononuclear cell (PBMC) samples by built-in MAST package and Wilcoxon rank-sum test, respectively. Single-cell trajectory analysis for single-cell RNA expression profile will be implemented by Monocle 3 to discover the transitions of cell states in the blood over the course of treatment.
Psuedotime gene trajectory | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Will be assessed by multiplex immunofluorescence. Cell classifications based on panel design will be created for all cell objects detected in whole slide images of tissues. Tissue segmentation for tumor and stroma areas will be created. Densities of cell classifications within whole tissue, tumor areas, and stroma areas will be calculated. Neighborhood analysis, based off 25micron radius, will be examined using Cytomap to identify patterns of cell-cell interactions within tissues. All quantitative image analysis data between pre-treatment and post-treatment samples will be compared in the context of clinical response to CDK4/6i by Wilcoxon rank-sum tests.
Cells per mm^2 tissue | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Will be assessed by multiplex immunofluorescence. Cell classifications based on panel design will be created for all cell objects detected in whole slide images of tissues. Tissue segmentation for tumor and stroma areas will be created. Densities of cell classifications within whole tissue, tumor areas, and stroma areas will be calculated. Neighborhood analysis, based off 25micron radius, will be examined using Cytomap to identify patterns of cell-cell interactions within tissues. All quantitative image analysis data between pre-treatment and post-treatment samples will be compared in the context of clinical response to CDK4/6i by Wilcoxon rank-sum tests.
Cells per mm^2 cancer island | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Will be assessed by multiplex immunofluorescence. Cell classifications based on panel design will be created for all cell objects detected in whole slide images of tissues. Tissue segmentation for tumor and stroma areas will be created. Densities of cell classifications within whole tissue, tumor areas, and stroma areas will be calculated. Neighborhood analysis, based off 25micron radius, will be examined using Cytomap to identify patterns of cell-cell interactions within tissues. All quantitative image analysis data between pre-treatment and post-treatment samples will be compared in the context of clinical response to CDK4/6i by Wilcoxon rank-sum tests.
Average cell-cell distances (within neighborhood) | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Will be assessed by multiplex immunofluorescence. Cell classifications based on panel design will be created for all cell objects detected in whole slide images of tissues. Tissue segmentation for tumor and stroma areas will be created. Densities of cell classifications within whole tissue, tumor areas, and stroma areas will be calculated. Neighborhood analysis, based off 25micron radius, will be examined using Cytomap to identify patterns of cell-cell interactions within tissues. All quantitative image analysis data between pre-treatment and post-treatment samples will be compared in the context of clinical response to CDK4/6i by Wilcoxon rank-sum tests.
Cells per mm^2 stroma | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Will be assessed by multiplex immunofluorescence. Cell classifications based on panel design will be created for all cell objects detected in whole slide images of tissues. Tissue segmentation for tumor and stroma areas will be created. Densities of cell classifications within whole tissue, tumor areas, and stroma areas will be calculated. Neighborhood analysis, based off 25micron radius, will be examined using Cytomap to identify patterns of cell-cell interactions within tissues. All quantitative image analysis data between pre-treatment and post-treatment samples will be compared in the context of clinical response to CDK4/6i by Wilcoxon rank-sum tests.
Number of core cells with cell(s) in neighborhood | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Will be assessed by multiplex immunofluorescence. Cell classifications based on panel design will be created for all cell objects detected in whole slide images of tissues. Tissue segmentation for tumor and stroma areas will be created. Densities of cell classifications within whole tissue, tumor areas, and stroma areas will be calculated. Neighborhood analysis, based off 25micron radius, will be examined using Cytomap to identify patterns of cell-cell interactions within tissues. All quantitative image analysis data between pre-treatment and post-treatment samples will be compared in the context of clinical response to CDK4/6i by Wilcoxon rank-sum tests.
Number of spatial clusters | From date of initiation of CDK4/6 inhibitor (either ribociclib or palbociclib) to disease progression (clinical or imaging), or, up to a maximum of 5 years
  Will be assessed by multiplex immunofluorescence. Cell classifications based on panel design will be created for all cell objects detected in whole slide images of tissues. Tissue segmentation for tumor and stroma areas will be created. Densities of cell classifications within whole tissue, tumor areas, and stroma areas will be calculated. Neighborhood analysis, based off 25micron radius, will be examined using Cytomap to identify patterns of cell-cell interactions within tissues. All quantitative image analysis data between pre-treatment and post-treatment samples will be compared in the context of clinical response to CDK4/6i by Wilcoxon rank-sum tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yuan, Principal Investigator — City of Hope Medical Center